CLINICAL TRIAL: NCT00705900
Title: A Randomized, Single-Blind, Active Control, 18-Week Study to Evaluate the Safety and Efficacy of A New Twice-Daily, Topically Applied LCD Solution vs. Calcipotriol Cream for the Treatment of Adult Subjects With Moderate Plaque Psoriasis
Brief Title: LCD Solution Versus Calcipotriol Cream in the Treatment of Moderate Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoStrata Company, Inc. (Industry)
Responsible Party: Alexandra B. Kimball, MD, Massachusettes General Hospital / Brigham Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-LCDPOP
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Plaque Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): LCD Solution: 2 applications / day
  Interventions: Drug: LCD
- 2 (Active Comparator): Calcipotriol cream: 2 applications / day
  Interventions: Drug: calcipotriol

INTERVENTIONS:
Drug: LCD — 2 applications / day for 12 weeks
  Arms: 1
Drug: calcipotriol — 2 applications / day for 12 weeks
  Other Names: Dovonex Cream (50 mcg/g 0.005%)
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of a new topical LCD solution and a commercially available calcipotriol (Vitamin D) cream in reducing the symptoms of plaque psoriasis and improving the quality of life in adults.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able and willing to provide written informed consent
* diagnosed with chronic plaque psoriasis
* 3% to 15% body surface area involved
* in good general health

Exclusion Criteria:

* other current treatments for psoriasis
* renal or liver dysfunction
* pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Difference in percent reduction in Psoriasis Area and Severity Index (PASI) Scores between treatment arms | 12 weeks of treatment

SECONDARY OUTCOMES:
Changes in PLASI, PEASI, Physician Global Assessment (PGA), Pruritus, and Dermatology Life Quality Index (DLQI) Scores between treatment arms | Week 12 and Week 18

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, Principal Investigator — Massachusettes General Hospital / Brigham Women's Hospital
Locations (1):
- Mass General Hospital: Clinical Unit for Research Trials in Skin, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Alora-Palli MB, Brouda I, Green B, Kimball AB. A cost-effectiveness comparison of liquor carbonis distillate solution and calcipotriol cream in the treatment of moderate chronic plaque psoriasis. Arch Dermatol. 2010 Aug;146(8):919-22. doi: 10.1001/archdermatol.2010.167. No abstract available. PMID 20713833
- [Derived] Alora-Palli MB, Perkins AC, Van Cott A, Kimball AB. Efficacy and tolerability of a cosmetically acceptable coal tar solution in the treatment of moderate plaque psoriasis: a controlled comparison with calcipotriene (calcipotriol) cream. Am J Clin Dermatol. 2010;11(4):275-83. doi: 10.2165/11530380-000000000-00000. PMID 20513160